CLINICAL TRIAL: NCT04990492
Title: Interactive Voice Based Administration of the GAD 7
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oklahoma State University Center for Health Sciences (Other)
Collaborators: Oral Roberts University (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021029
Record Dates: First submitted 2021-07-06; First posted 2021-08-04 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: General Anxiety Disorder
MeSH Terms: conditions — Generalized Anxiety Disorder

STUDY DESIGN:
Intervention Model Description: This study will be a repeated measure, mixed methods design (i.e., it will contain both qualitative and quantitative components). Newly admitted patients will be asked to complete the questionnaires (i.e., GAD 7 and the UEQ) at two different time points (i.e., Baseline and 1-month follow-up). In order to reduce or control for order effects, the procedure will be counterbalanced.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paper Baseline (Experimental): Half of the participants will complete the GAD 7 in the traditional paper format at their first appointment. At their second appointment 1-month later, they will complete the GAD 7 on the Mirror device equipped with Amazon Alexa.
  Interventions: Diagnostic Test: Paper GAD 7; Diagnostic Test: Voice Administered GAD 7
- Alexa Baseline (Experimental): The other half of the participants will complete the GAD 7 on the Mirror device equipped with Amazon in the traditional paper format at their first appointment. At their second appointment 1-month later, they will complete the GAD 7 in the traditional paper format.
  Interventions: Diagnostic Test: Paper GAD 7; Diagnostic Test: Voice Administered GAD 7

INTERVENTIONS:
Diagnostic Test: Paper GAD 7 — The paper based GAD 7 that is commonly accepted at clinics
  Other Names: Clinically Accepted Paper GAD 7
Diagnostic Test: Voice Administered GAD 7 — This is the voice based GAD 7 that is administered through a Mirror device equipped with Amazon Alexa software.
  Other Names: Alexa GAD 7; Mirror GAD 7

SUMMARY:
This study investigates a new delivery method for the General Anxiety Disorder - 7 (GAD 7), a clinically accepted tool for diagnosing general anxiety disorder. The new tool records auditory responses to the assessment and the study will examine if the instrument is effective at capturing participant depression levels. If proven effective, future studies may investigate if the new format can be used to improve at home clinical care.

DETAILED DESCRIPTION:
This study is an investigation of the construct validity and user experience of a new delivery system for the General Anxiety Disorder - 7 (GAD 7), a clinically accepted tool for diagnosing general anxiety disorder. The purpose of the study is to examine if the new delivery system of the GAD 7 is effective at capturing participant anxiety levels and to assess the differences of usability between the paper and voice administered versions. The voice administered version uses a Mirror device, which is similar to a smart television with a mirror interface. The device records auditory responses to the GAD 7 through Amazon Alexa. The investigators will be comparing the responses on the new device to those given on the clinically established paper format. If proven effective at capturing depression levels of patients, future studies may investigate if the new format can be used to improve at home clinical care.

ELIGIBILITY:
Inclusion Criteria::

* Newly admitted patients to the Oklahoma State University Behavioral Medicine Clinic

Exclusion Criteria:

* Vulnerable populations, such as children (i.e., minors or individuals under the legal age of consent) and individuals who are incarcerated (i.e., prisoners), will be excluded.
* Individuals who are not their own guardian (i.e., those suffering from severe disabilities) will also be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-06-10 (Actual); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-06-15 (Estimated)

PRIMARY OUTCOMES:
GAD 7 Diagnostic Scores | Five minutes
  Scores from the self administered assessment for general anxiety disorder
User Experience Questionnaire | Five minutes
  Likert based questionnaire on user experience

SECONDARY OUTCOMES:
Patient's Qualitative Responses | One minute
  Comments from patient on usability of the device

CONTACTS AND LOCATIONS:
Overall Officials: Jason Beaman, D.O., Principal Investigator — Oklahoma State University Center for Health Sciences
Locations (1):
- OSU Behavioral Health Clinic, Tulsa, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No
Aggregate data and findings will be posted on ClinicalTrials.gov.

DOCUMENTS (1):
  • Informed Consent Form (2021-04-22): https://cdn.clinicaltrials.gov/large-docs/92/NCT04990492/ICF_000.pdf